CLINICAL TRIAL: NCT03033602
Title: Brief Treatment for PTSD: Enhancing Retention and Engagement
Brief Title: Brief Treatment for Posttraumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston VA Research Institute, Inc. (Other)
Collaborators: University of Texas (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81WH-15-1-0391
Record Dates: First submitted 2016-12-02; First posted 2017-01-27 (Estimated); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2022-07

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Written exposure therapy (Experimental): 5 sessions of imaginal exposure therapy.
  Interventions: Behavioral: written exposure therapy
- CPT, cognitive only (Active Comparator): 12 sessions of cognitive therapy.
  Interventions: Behavioral: CPT, cognitive only

INTERVENTIONS:
Behavioral: written exposure therapy — five sessions of writing about traumatic experience.
  Other Names: WET
  Arms: Written exposure therapy
Behavioral: CPT, cognitive only — 12 sessions of cognitive therapy related to traumatic experience.
  Other Names: CPT-C
  Arms: CPT, cognitive only

SUMMARY:
The primary goal of this study is to examine whether a brief treatment approach for PTSD is equally efficacious in the treatment of active duty service members relative to a first line treatment approach that requires much greater treatment dose.

DETAILED DESCRIPTION:
The goal of this randomized clinical trial is to investigate if a brief, written intervention for posttraumatic stress disorder (PTSD), Written Exposure Therapy (WET), is non-inferior compared to an evidenced-based behavioral therapy, Cognitive Processing Therapy-Cognition only (CPT-C), in the treatment of PTSD in active duty military men and women with a diagnosis of PTSD who have deployed in support of a post-9/11. The primary study outcome is change in symptom severity as assessed by the Clinician Administered PTSD Scale for Diagnostic and Statistical Manual-5 edition (CAPS-5). Independent assessors evaluated participants using the CAPS-5 at baseline, 10-, 20-, and 30-week after the first treatment session.

ELIGIBILITY:
Inclusion Criteria:

* Male and female active duty military personnel who have deployed in support of a post-9/11 conflict seeking treatment for PTSD
* Diagnosis of PTSD
* Ability to speak, read and write English
* Not currently engaged in psychosocial treatment for PTSD
* Individuals taking psychotropic medications agree to work with their prescriber to remain on stable doses of any prescribed psychotropic medications for the duration of the intervention and through the first follow-up assessment as much as possible and as medically indicated.

Exclusion Criteria:

* Current suicide or homicide risk meriting crisis intervention
* Active psychosis
* Moderate to severe brain damage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2015-07-20 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Sloan, Ph.D., Principal Investigator — Boston VA Research Institute, Inc.
Locations (2):
- United States (2):
  - Ft. Hood, Killeen, Texas
  - University of Texas Health Science Center, San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon written request to the PI.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 12 months after publication of the primary outcomes.
Access Criteria: Written request to the PI describing rationale for why data is needed and what will be done with data.

REFERENCES:
- [Background] Sloan DM, Marx BP, Resick PA, Young-McCaughan S, Dondanville KA, Straud CL, Mintz J, Litz BT, Peterson AL; STRONG STAR Consortium. Effect of Written Exposure Therapy vs Cognitive Processing Therapy on Increasing Treatment Efficiency Among Military Service Members With Posttraumatic Stress Disorder: A Randomized Noninferiority Trial. JAMA Netw Open. 2022 Jan 4;5(1):e2140911. doi: 10.1001/jamanetworkopen.2021.40911. PMID 35015065
- [Background] Sloan DM, Marx BP, Resick PA, Young-McCaughan S, Dondanville KA, Mintz J, Litz BT, Peterson AL; STRONG STAR Consortium. Study design comparing written exposure therapy to cognitive processing therapy for PTSD among military service members: A noninferiority trial. Contemp Clin Trials Commun. 2019 Dec 10;17:100507. doi: 10.1016/j.conctc.2019.100507. eCollection 2020 Mar. PMID 31890987

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Written Exposure Therapy | CPT, Cognitive Only
Started | 85 | 84
Completed (completed treatment) | 65 | 47
Not Completed | 20 | 37
Not completed — Withdrawal by Subject | 11 | 21
Not completed — discontinued for medical reason or decision by study team | 9 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Written Exposure Therapy | CPT, Cognitive Only | Total
Number analyzed (Participants) | 85 | 84 | 169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 85 | 84 | 169
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.98 (6.86) | 33.32 (8.22) | 33.65 (8.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 69 | 67 | 136
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 3 | 4 | 7
  Black or African American | 28 | 29 | 57
  White | 33 | 26 | 59
  More than one race | 20 | 24 | 44
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 85 | 84 | 169

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale, 5 (CAPS-5)
Description: The CAPS-5 is a semi-structured interview for assessment of PTSD according to DSM-5 diagnostic criteria. The measure assesses PTSD according to the 20 symptoms of DSM-5, as well as impairment. A total score is calculated as well as whether PTSD diagnosis is met. Scores can range from 0-80, with higher scores representing greater symptom severity. For this study, the CAPS-5 total score was used as the primary outcome measure.
Time Frame: Change from baseline to 10-, 20-, 30-weeks post first treatment session
Population: Non-inferiority margin
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Written Exposure Therapy | CPT, Cognitive Only
Number analyzed (Participants) | 85 | 84
score on a scale
  10-week assessment | 31.55 (1.13) | 25.12 (1.40)
  20 week assessment | 29.59 (1.45) | 25.41 (1.49)
  30 week assessment | 27.77 (1.61) | 24.97 (1.68)

ADVERSE EVENTS:
Time Frame: 6 months.
Arm/Group | Written Exposure Therapy | CPT, Cognitive Only
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/84
Serious Adverse Events (participants affected / at risk) | 1/85 | 1/84
Other Adverse Events (participants affected / at risk) | 6/85 | 7/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Written Exposure Therapy (N=85) | CPT, Cognitive Only (N=84)
psychiatric hospitalization (Psychiatric disorders) | 1 (1) | 1 (1) — admitted to psychiatric unit due to suicidality
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Written Exposure Therapy (N=85) | CPT, Cognitive Only (N=84)
increase in anxiety symptoms (Psychiatric disorders) | 6 (6) | 7 (7)

LIMITATIONS AND CAVEATS:
Participants who dropped out prematurely of treatment were less likely to return for subsequent assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/02/NCT03033602/Prot_SAP_000.pdf